CLINICAL TRIAL: NCT02954224
Title: Prevention Of Delirium in Elderly With Obstructive Sleep Apnea (PODESA)
Acronym: PODESA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jean Wong, Dr., University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014-0122-B
Record Dates: First submitted 2016-09-23; First posted 2016-11-03 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Sleep Apnea
Keywords: sleep apnea, delirium
MeSH Terms: conditions — Sleep Apnea Syndromes; Delirium | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CPAP therapy arm (Experimental): Auto-titrating Continuous Positive Airway Pressure (CPAP)) treatment will be given on postoperative days 1, 2, and 3.
  Interventions: Other: CPAP treatment
- Control arm (No Intervention): no auto-titrating CPAP, standard care

INTERVENTIONS:
Other: CPAP treatment — Patients who are randomized to auto-titrating CPAP will use an auto CPAP device on postoperative days 1, 2, and 3
  Arms: CPAP therapy arm

SUMMARY:
Delirium is a common complication in elderly patients following surgery. Patients who develop delirium after surgery are at increased risk for serious complications, and even death.This multi-centre randomized controlled trial will enroll elderly patients scheduled for elective hip/knee replacement surgery.The objective of this trial is to identify obstructive sleep apnea using ApneaLink Air and to determine whether auto-titrating CPAP treatment of obstructive sleep apnea will decrease the incidence of post-operative delirium in elderly patients undergoing elective hip and knee replacement surgery.

DETAILED DESCRIPTION:
Delirium is an acute and fluctuating change in cognitive function, characterized by poor attention and disorganized thinking. Recent studies show that patients with obstructive sleep apnea (OSA) - a sleep disorder characterized by repeated episodes of complete or partial blockage of the upper airway - are at greater risk to develop delirium. It is estimated that 43% of men and 27% of women aged 50-70 years old have OSA. Elderly individuals with this condition are often undiagnosed. Unrecognized OSA may be a treatable cause of postoperative delirium. However, timely access to polysomnography is usually not possible prior to surgery. This multi-centre randomized controlled trial will enroll elderly patients scheduled for elective hip/knee replacement surgery. All participants who have given the consent to participate will be assessed risks of OSA and comorbidity by 3 basic questionnaires- STOP-Bang, Epworth Sleepiness Scale and Charlson Comorbidity index, Cognitive level assess by Mini-Cog and baseline delirium assessment by CAM. STOP-Bang questionnaire is the validated questionnaire to screen the patients for OSA. Score of 3 or higher has sensitivity of detecting OSA of 93% and 100% for moderate and severe OSA respectively. If participant has STOP-Bang score 3 or higher will have a home sleep study with the ApneaLink Air and overnight oximetry. Patients identified to have OSA(AHI ≥10/h) will be randomized to 1) Auto-titrating continuous positive airway pressure (CPAP) applied 1-3 nights before surgery (if possible) and during day/night sleep for 72 hrs after surgery or 2) Control group - routine care. All patients will be evaluated for delirium for 72h after surgery.

ELIGIBILITY:
Inclusion criteria

* Age more than 60 years, Scheduled for elective hip or knee replacement surgery at least 4 working days after the preadmission clinic visit
* Possess cognitive and physical capability necessary to comprehend and complete the study questionnaires
* Proficient in English, reading level at Grade 6 (patient or accompanying person),
* Be accessible for follow-up via telephone, or via the Internet, Ability to provide informed consent

Exclusion criteria

* Conditions potentially interfering with comprehension and delivery of informed consent , Schizophrenia, anxiety disorders, poorly controlled depression, multiple psychiatric disorders
* Active psychosis within the last 3 months
* Current use of antipsychotic medication
* Dementia, and/or clinically significant neurological disorder (stroke, epilepsy, brain tumors, Parkinson's Disease etc.)
* History of drug or alcohol dependence or abuse within last 3 months
* Surgery that is two-staged involving more than one surgical procedure to be performed within the same hospitalization period
* Emergency surgery when preoperative testing is not possible
* Patients with prior diagnosis of sleep-related breathing disorder with CPAP treatment
* Patients who may have had sleep studies earlier may be included, if they have been lost to follow-up by a sleep physician, are not on treatment or are non-compliant to treatment (mean CPAP nightly use <4 hours, or median nightly CPAP use <50% of total sleep time),Severe tracheal or lung disease,Contraindication to CPAP face-mask, Central Sleep Apnea, Significant Cardiac disease(New York Heart Association Functional Class III and IV Severe Valvular Heart Disease, Dilated Cardiomyopathy, Implanted Cardiac Pacemaker, unstable angina)
* bMyocardial Infarction or Cardiac Surgery or Percutaneous coronary interventions within 3 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
postoperative delirium | 2 MONTHS
  The primary outcome is the incidence of postoperative delirium.

SECONDARY OUTCOMES:
Length of Hospital Stay | Depending on post operative recovery(2 days-2 months)
  This parameter depends on post operative recovery
Time to ambulate | 1 week to 2 months
  This parameter depending on lots of factors( eg; physiotherapy, weight, attitudes, other medical conditions ect...)
Perioperative Complications | 10-14 days
  Post operative complications include ICU admissions, hypoxia, re-intubation, Myocardial Infarctions, Wound Infections, Deep Vein Thrombosis, Pneumonia, Sepsis, Urinary Tract Infection, Stroke, etc..)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wong, MD, Principal Investigator — University Health Network, Toronto
Locations (3):
- Canada (3):
  - Sunnybrook Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong J, Doherty HR, Singh M, Choi S, Siddiqui N, Lam D, Liyanage N, Tomlinson G, Chung F. The prevention of delirium in elderly surgical patients with obstructive sleep apnea (PODESA): a randomized controlled trial. BMC Anesthesiol. 2022 Sep 14;22(1):290. doi: 10.1186/s12871-022-01831-1. PMID 36104664
- [Derived] Wong J, Lam D, Choi S, Singh M, Siddiqui N, Sockalingam S, Chung F. The prevention of delirium in elderly with obstructive sleep apnea (PODESA) study: protocol for a multi-centre prospective randomized, controlled trial. BMC Anesthesiol. 2018 Jan 3;18(1):1. doi: 10.1186/s12871-017-0465-5. PMID 29298664